CLINICAL TRIAL: NCT02847819
Title: Pre and Post-operative Evaluation of Vocal Cord Movement in Patients Undergoing Thyroid Surgery by Airway Ultrasound Scanning.
Brief Title: Vocal Cord Movement Assessment Using Airway Ultrasound.
Status: Completed | Type: Observational
Sponsor: Rajiv Gandhi Cancer Institute & Research Center, India (Other)
Responsible Party: Principal Investigator, Amit Kumar Mittal, Doctor, Rajiv Gandhi Cancer Institute & Research Center, India
Other Study IDs: RGCI ID: 506/AN/AKM-04
Record Dates: First submitted 2016-07-25; First posted 2016-07-28 (Estimated); Last update posted 2020-06-18 (Actual); Status verified 2017-04

CONDITIONS: Vocal Cord Movement Assessment by Airway Ultrasound

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Vocal cords movement assessment by airway USG.: Preoperatively patients undergoing thyroid surgery will be scanned by airway ultrasound and graded for vocal cord movement, the same group of patients will be again scanned and graded by airway ultrasound at 4th post operative hours.
  Interventions: Device: airway ultrasound for vocal cords movement assessment.

INTERVENTIONS:
Device: airway ultrasound for vocal cords movement assessment. — Glottic aperture will be scanned using 7.5 megahertz (MHz) linear transducer portable ultrasound machine. after getting the best acoustic window, true, false vocal cords arytenoid movements will be visualized. Individual cord will be focused and doppler velocity will be measured for both the cords.

SUMMARY:
Total of 100 patients are included in this is a prospective observational study to evaluate the role of airway ultrasound (USG) in assessing vocal cord mobility in patients undergoing thyroid surgery. patients will be scanned preoperatively by airway ultrasound which will be compared to post operative ultrasound scans.

DETAILED DESCRIPTION:
All 100 patients between age groups of 15-70 years, will be scanned pre-operatively to see vocal cord mobility as a reference value. A proper acoustic window is mandatory for optimal visualization of laryngeal structures. Visibility of false vocal cords, true vocal cords and arytenoids will be given one point each for one side, maximal score will be 6. According to points the acoustic window scoring for glottis aperture will be graded as fair, when both false vocal cords are visible (score1-2), along with false cord when both arytenoids are visible scored good (score3-4) and if single or both true vocal cords are visible then scored as very good(score5-6). After the surgery the same patient will be scanned again for vocal cord mobility at 4hours of extubation . Any change in mobility will be recorded. If any change will be observed, direct laryngoscopy (DL) will be done to confirm the diagnosis. Any complication in the post-operative period will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing thyroid surgery between specified age limits.

Exclusion Criteria:

* Retro sternal goiters.

Ages: 17 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients undergoing thyroid surgery.
Sampling Method: Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2016-07-02 (Actual); Primary Completion 2017-08-17 (Actual); Study Completion 2017-08-25 (Actual)

PRIMARY OUTCOMES:
Objective confirmation of vocal cords movement | pre operatively and at 4 hours after extubation

SECONDARY OUTCOMES:
Comparison of preoperative doppler velocity with post operative doppler velocity. | At 4 hours after extubation.

CONTACTS AND LOCATIONS:
Overall Officials: Mamta Dubey, M.D, Principal Investigator — Rajiv Gandhi Cancer Institute & Research Centre, Rohini; New Delhi: India 110085.
Locations (1):
- Rajiv Gandhi Cancer Institute & Research center, Delhi, New Delhi, India

REFERENCES:
- [Derived] Dubey M, Mittal AK, Jaipuria J, Arora M, Dewan AK, Pahade A. Functional analysis of vocal folds by transcutaneous laryngeal ultrasonography in patients undergoing thyroidectomy. Acta Anaesthesiol Scand. 2019 Feb;63(2):178-186. doi: 10.1111/aas.13234. Epub 2018 Aug 5. PMID 30079464